CLINICAL TRIAL: NCT04564833
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Effect of RBT-1 on Preconditioning Response Biomarkers in Subjects Undergoing Coronary Artery Bypass Graft (CABG) and/or Cardiac Valve Surgery (The START Study)
Brief Title: Effect of RBT-1 on Preconditioning Response Biomarkers in Subjects Undergoing CABG and/or Cardiac Valve Surgery
Acronym: START
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renibus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REN-004
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Results first posted 2024-01-16 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: AKI

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1:1 to low dose RBT-1, high dose RBT-1, and placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose RBT-1 (Experimental): Single IV infusion prior to cardiac surgery
  Interventions: Drug: Low Dose RBT-1
- High Dose RBT-1 (Experimental): Single IV infusion prior to cardiac surgery
  Interventions: Drug: High Dose RBT-1
- Placebo (Placebo Comparator): Single IV infusion prior to cardiac surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low Dose RBT-1 — intravenous administration
  Arms: Low Dose RBT-1
Drug: High Dose RBT-1 — intravenous administration
  Arms: High Dose RBT-1
Drug: Placebo — intravenous administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of RBT-1 (stannous protoporphyrin [SnPP]/iron sucrose [FeS]) on preconditioning response biomarkers in subjects who are at risk for AKI following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years of age at Screening.
2. Able and willing to comply with all study procedures.
3. Stable kidney function per Investigator assessment and no known episodes of AKI during the preceding 4 weeks.
4. Scheduled to undergo non-emergent coronary and/or valve surgery(ies) requiring cardiopulmonary bypass, including:

   * CABG alone;
   * Combined CABG surgery/repair of 1 or more cardiac valves;
   * Cardiac valve(s) replacement or repair alone.
5. Females and males of childbearing potential must agree to use 2 forms of contraception, with at least 1 being a barrier method, or abstain from sexual activity for 30 days following study drug administration.
6. Male subjects must agree not to donate or sell sperm for 30 days following study drug administration.

Exclusion Criteria:

1. Presence of AKI (KDIGO criteria) at the time of Screening.
2. Surgery to be performed without cardiopulmonary bypass.
3. Surgery to be performed under conditions of circulatory arrest or hypothermia with rectal temperature <28°C (82.4°F).
4. eGFR ≤20 mL/min/1.73m2 or need for dialysis.
5. Surgery for aortic dissection or to correct a major congenital heart defect.
6. Administration of iodinated contrast media within 24 hours prior to cardiac surgery or evidence of contrast-induced nephropathy prior to cardiac surgery.
7. Cardiogenic shock or hemodynamic instability within the 24 hours prior to surgery and requirement for inotropes or vasopressors or other mechanical devices, such as intra-aortic balloon counter-pulsation.
8. Requirement for any of the following within 7 days prior to cardiac surgery:

   * Defibrillator or permanent pacemaker;
   * Mechanical ventilation;
   * Intra-aortic balloon counter-pulsation;
   * Left ventricular assist device;
   * Other forms of mechanical circulatory support.
9. Known history of cancer within the past 2 years, except for carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin.
10. Known or suspected sepsis at time of Screening or confirmed or treated endocarditis within 30 days prior to cardiac surgery.
11. Other current active infection requiring systemic antibiotic treatment.
12. Inadequate hepatic function, defined as total bilirubin or alanine aminotransferase or aspartate aminotransferase >2X the upper limit of normal at time of Screening or Child Pugh Class C liver disease or higher.
13. Any congenital coagulation disorder.
14. Asplenia (anatomic or functional).
15. History of photosensitivity or active skin disease that, in the opinion of the Investigator, could be worsened by RBT-1.
16. Known hypersensitivity or previous anaphylaxis to SnPP or any tin-based product.
17. Serum ferritin >500 ng/mL or those who have received IV iron within 28 days of Screening.
18. Pregnancy or lactation.
19. Treatment with an investigational drug or participation in an interventional study within 30 days prior to administration of study drug.
20. In the opinion of the Investigator, any disease processes or confounding variables that would inappropriately alter the outcome of the study.
21. Inability to comply with the requirements of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2023-02-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (18):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Keck Hospital of USC, Los Angeles, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Stanford University Medical Center, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Health Research Institute, Inc., Washington D.C., District of Columbia
  - University of Chicago Hospital Anesthesia and Critical Care, Chicago, Illinois
  - Indiana University Health Southern Indiana, Bloomington, Indiana
  - Lutheran Medical Group, Fort Wayne, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - McLaren Greater Lansing, Lansing, Michigan
  - MyMichigan Medical Center, Midland, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - New York Presbyterian-Queens, Flushing, New York
  - Columbia University Irving Medical Center, New York, New York
  - Rochester General Hospital Center for Clinical Research, Rochester, New York
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Australia (4):
  - Gold Cost University Hospital & Health Services, Southport, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Canada (3):
  - St-John Regional Hospital, Saint John, New Brunswick
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lamy A, Chertow GM, Jessen M, Collar A, Brown CD, Mack CA, Marzouk M, Scavo V, Washburn TB, Savage D, Smith J, Bennetts J, Assi R, Shults C, Arghami A, Butler J, Devereaux PJ, Zager R, Wang C, Snapinn S, Browne A, Rodriguez J, Ruiz S, Singh B; of START Investigators. Effects of RBT-1 on preconditioning response biomarkers in patients undergoing coronary artery bypass graft or heart valve surgery: a multicentre, double-blind, randomised, placebo-controlled phase 2 trial. EClinicalMedicine. 2024 Jan 8;68:102364. doi: 10.1016/j.eclinm.2023.102364. eCollection 2024 Feb. PMID 38586479
- See also: Effects of RBT-1 on preconditioning response biomarkers in patients undergoing coronary artery bypass graft or heart valve surgery: a multicentre, double-blind, randomised, placebo-controlled phase 2 trial — https://pubmed.ncbi.nlm.nih.gov/38586479/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants were excluded after signing informed consent (11 did not meet eligibility criteria, 5 withdrew consent prior to treatment, 1 had surgery changed to another location)
Groups:
- High Dose RBT-1: Single IV infusion of high dose RBT-1 within 1-2 days prior to scheduled cardiac surgery
- Low Dose RBT-1: Single IV infusion of low dose RBT-1 within 1-2 days prior to scheduled cardiac surgery
- Placebo: Single IV infusion of placebo within 1-2 days prior to scheduled cardiac surgery
Period: Overall Study
Arm/Group | High Dose RBT-1 | Low Dose RBT-1 | Placebo
Started | 46 | 45 | 44
Completed | 46 | 45 | 44
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose RBT-1 | Low Dose RBT-1 | Placebo | Total
Number analyzed (Participants) | 46 | 45 | 44 | 135
Age, Continuous [Mean (Full Range); unit: years] | 66.04 [37 to 86] | 63.87 [46 to 82] | 65.70 [19 to 81] | 65.21 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 12 | 33
  Male | 36 | 34 | 32 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 45 | 41 | 43 | 129
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 1 | 4
  Black or African American | 2 | 4 | 2 | 8
  White | 41 | 38 | 41 | 120
  Other | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 9 | 10 | 27
  United States | 33 | 32 | 31 | 96
  Australia | 5 | 4 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Efficacy of RBT-1 in Generating a Preconditioning Response as Measured by a Composite of Biomarkers
Description: Composite of the geometric mean of the ratios of the maximum PreOp value over Baseline for plasma heme oxygenase-1 (HO-1), ferritin, and interleukin-10 (IL-10)
Time Frame: Baseline through Pre-Surgery
Population: Values were missing from 3 subjects in the low dose RBT-1 treatment group.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: composite ratio
Groups:
- High Dose RBT-1; Low Dose RBT-1; Placebo: Intention-To-Treat (ITT) Population - all subjects who had biomarker assessments at Baseline and prior to surgery
Arm/Group | High Dose RBT-1 | Low Dose RBT-1 | Placebo
Number analyzed (Participants) | 46 | 42 | 44
composite ratio | 3.60 [3.10 to 4.18] | 2.63 [2.25 to 3.07] | 1.00 [0.86 to 1.17]
Statistical Analysis 1: Comparison: High Dose RBT-1 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Low Dose RBT-1 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA

2. Secondary Outcome: Change in Renal Tubular Injury Biomarkers
Description: Geometric mean of the ratios of the maximum PostOp value over Baseline for urine KIM-1, NGAL, and cystatin C.
Time Frame: Baseline through Day 3 post-cardiac surgery
Population: Biomarker samples were missing from 2 subjects in the Low Dose RBT-1 group and 1 subject in the Placebo group.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Composite ratio
Groups:
- High Dose RBT-1; Low Dose RBT-1; Placebo: Modified Intention-To-Treat (MITT) Population - all subjects in the ITT population who underwent cardiac surgery without delay
Arm/Group | High Dose RBT-1 | Low Dose RBT-1 | Placebo
Number analyzed (Participants) | 41 | 37 | 40
Composite ratio | 7.89 [5.09 to 12.23] | 10.84 [6.92 to 16.98] | 6.10 [3.96 to 9.39]
Statistical Analysis 1: Comparison: High Dose RBT-1 vs Placebo; Test type: Superiority; p = 0.3954, ANCOVA
Statistical Analysis 2: Comparison: Low Dose RBT-1 vs Placebo; Test type: Superiority; p = 0.0682, ANCOVA

3. Secondary Outcome: Number of Subjects With Reduction in Urine Output
Description: Documented AE of sustained reduction in urine output, oliguria, or anuria post-cardiac surgery through Day 5
Time Frame: Baseline through post-cardiac surgery through Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose RBT-1 | Low Dose RBT-1 | Placebo
Number analyzed (Participants) | 41 | 39 | 41
Participants | 2 | 2 | 4
Statistical Analysis 1: Comparison: High Dose RBT-1 vs Placebo; Test type: Superiority; p = 0.6755, Fisher Exact
Statistical Analysis 2: Comparison: Low Dose RBT-1 vs Placebo; Test type: Superiority; p = 0.6758, Fisher Exact

4. Secondary Outcome: Number of Subjects With Acute Kidney Injury (AKI)
Description: AKI is defined using the KDIGO criteria (ie, an absolute increase in serum creatinine of ≥1.5 × Baseline; or documented AE of sustained reduction in urine output, oliguria, or anuria; or initiation of dialysis).
Time Frame: Baseline through Day 5 post-cardiac surgery
Measure: Count of Participants; unit: Participants
Arm/Group | High Dose RBT-1 | Low Dose RBT-1 | Placebo
Number analyzed (Participants) | 41 | 39 | 41
Participants | 7 | 7 | 8
Statistical Analysis 1: Comparison: High Dose RBT-1 vs Placebo; Test type: Superiority; p > 0.9999, Fisher Exact
Statistical Analysis 2: Comparison: Low Dose RBT-1 vs Placebo; Test type: Superiority; p > 0.9999, Fisher Exact

ADVERSE EVENTS:
Time Frame: An average of 90 days from the start of dosing
Arm/Group | High Dose RBT-1 | Low Dose RBT-1 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/46 | 1/45 | 3/44
Serious Adverse Events (participants affected / at risk) | 22/46 | 13/45 | 18/44
Other Adverse Events (participants affected / at risk) | 42/46 | 40/45 | 40/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose RBT-1 (N=46) | Low Dose RBT-1 (N=45) | Placebo (N=44)
Blood loss anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 2
Cardiogenic shock (Cardiac disorders) | 1 | 2 | 1
Low cardiac output (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal ischemia (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1
Pneumonia pseudomonas (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1
Systemic candida (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post pericardiotomy syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Carbon dioxide increased (Investigations) | 1 | 0 | 0
Hypervolemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 1
Hypoglycemic seizure (Nervous system disorders) | 0 | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0 | 0
Device dislocation (Product Issues) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1
Hemorrhage (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | High Dose RBT-1 (N=46) | Low Dose RBT-1 (N=45) | Placebo (N=44)
Anemia (Blood and lymphatic system disorders) | 6 | 8 | 11
Blood loss anemia (Blood and lymphatic system disorders) | 1 | 4 | 4
Leukocytosis (Blood and lymphatic system disorders) | 4 | 3 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4 | 3
Atrial fibrillation (Cardiac disorders) | 10 | 10 | 16
Cardiomegaly (Cardiac disorders) | 2 | 3 | 2
Abdominal distention (Gastrointestinal disorders) | 1 | 0 | 3
Constipation (Gastrointestinal disorders) | 5 | 4 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 3
Nausea (Gastrointestinal disorders) | 14 | 9 | 9
Vomiting (Gastrointestinal disorders) | 0 | 2 | 3
Chest pain (General disorders) | 2 | 1 | 3
Generalized edema (General disorders) | 3 | 3 | 5
Edema (General disorders) | 2 | 2 | 4
Edema peripheral (General disorders) | 3 | 6 | 2
Pain (General disorders) | 1 | 1 | 5
Urinary tract infection (Infections and infestations) | 5 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 4 | 6 | 2
Procedural pain (Injury, poisoning and procedural complications) | 9 | 9 | 11
Breath sounds abnormal (Investigations) | 1 | 3 | 1
Urine output decreased (Investigations) | 6 | 4 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 5 | 5
Hypervolemia (Metabolism and nutrition disorders) | 5 | 4 | 9
Delirium (Psychiatric disorders) | 1 | 3 | 3
Hallucination (Psychiatric disorders) | 1 | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 5 | 5
Acute kidney injury (Renal and urinary disorders) | 3 | 7 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 8
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 10 | 6 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 3 | 2 | 0
Hypotension (Vascular disorders) | 12 | 11 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Center and Investigator shall not publish or present the Study results until after the first publication or presentation regarding the overall study is completed, such publication or presentation to be at the sole discretion of Sponsor, or eighteen (18) months from the completion date of the Study (as defined in 42 U.S.C. 282(j)(1)(A)(v)), whichever occurs first.

DOCUMENTS (2):
  • Study Protocol (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT04564833/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT04564833/SAP_001.pdf